CLINICAL TRIAL: NCT05664984
Title: The Effectiveness of Cognitive Rehabilitation Intervention With the Telerehabilitation Method for Amnestic Mild Cognitive Impairment: A Feasibility Randomized Controlled Trial
Brief Title: Effectiveness of Cognitive Rehabilitation for Amnestic Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Berkan Torpil, PhD, Associate professor, Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20/513
Record Dates: First submitted 2022-12-09; First posted 2022-12-27 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Mild Cognitive Impairment; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Intervention Model Description: single blind randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: The investigator who evaluated the cases was blinded from the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-face-to-face group (Experimental): Cognitive rehabilitation intervention was given face-to-face.
  Interventions: Behavioral: 1-face-to-face
- 2-tele rehabilitation group (Experimental): Cognitive rehabilitation intervention was given tele-rehabilitation method.
  Interventions: Behavioral: 2-tele rehabilitation

INTERVENTIONS:
Behavioral: 1-face-to-face — The cognitive rehabilitation intervention consists of 45-minute sessions, 2 days a week for 12 weeks. The same rehabilitation intervention program was applied to both groups by face-to-face or tele-rehabilitation method. The main purpose of the study is to see the effectiveness of cognitive rehabilitation intervention in the elderly with amnestic mild cognitive impairment and to compare the two methods.
  Other Names: Cognitive rehabilitation
  Arms: 1-face-to-face group
Behavioral: 2-tele rehabilitation — 2-tele rehabilitation
  Other Names: Cognitive rehabilitation
  Arms: 2-tele rehabilitation group

SUMMARY:
Different cognitive rehabilitation intervention methods have been developed for the treatment of cognitive dysfunctions seen in mild cognitive impairment (MCI). The aim of this study was to examine the effectiveness of cognitive rehabilitation intervention applied with the telerehabilitation method in elderly patients with amnestic-MCI.

Participants included in the study according to inclusion and exclusion criteria were randomly assigned to the telerehabilitation and face-to-face groups. A 12-week cognitive rehabilitation intervention was applied to both groups. Pre- and post-intervention cognitive skills of the participants were evaluated using the Loewenstein Occupational Therapy Cognitive Assessment-Geriatric (LOTCA-G).

DETAILED DESCRIPTION:
A single-blinded, feasibility randomized controlled trial (RCT) investigated changes in the cognitive functions of older adults with amnestic-MCI after CR interventions applied face-to-face and with telerehabilitation. The study was designed according to the CONSORT statement. Approval for the study was granted by the Local Ethics Committee. Written informed consent was obtained from all participants prior to the study.

The demographic characteristics of the participants were recorded, including age, sex, education level, and marital status. All participants underwent a cognitive function assessment using the Loewenstein Occupational Therapy Cognitive Assessment-Geriatric twice, once before the intervention and again after the 12-week intervention. All participants were assessed in occupational therapy clinical practice units.

Participants were randomized to either the Face-to-Face group (FF) or the Tele-rehabilitation group (TR) using a computer-generated randomization technique.

After the randomization, cognitive rehabilitation intervention for both methods consist of 45-minute twice a week for 12 weeks. All participants received the intervention individually.

ELIGIBILITY:
Inclusion Criteria:

* Age between 65 and 75 years
* Diagnosed with amnestic-MCI by medical doctors
* Access to technological equipment; and
* Ability to understand and follow verbal instructions.

Exclusion Criteria:

* Secondary chronic disease that may affect cognitive functioning;
* Auditory and visual problems that may affect rehabilitation implementation and communication; and
* Attendance of any rehabilitation program (physiotherapy, speech therapy, psychotherapy, etc.) during the study period.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 68 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
The Loewenstein Occupational Therapy Cognitive Assessment-Geriatric (LOTCA-G) | before the first session
  The LOTCA-G, which was created to evaluate cognitive functions in the elderly. This test evaluates 8 cognitive domains with 24 items: orientation, visual perception, spatial perception, motor praxis, visuomotor organization, thinking operations, attention/concentration, and memory. The items in each subtest are evaluated on an ordered scale from 1 to 4 (excluding the orientation items scored from 1 to 8). A higher test score indicates better cognitive performance. The LOTCA-G can differentiate healthy older adults from those with dementia and MCI. It is sensitive to dementia levels and identifies changes over time. The LOTCA-G was used to evaluate the effectiveness of cognitive rehabilitation intervention both face-to-face and with tele-rehabilitation method. It was planned to evaluate the effectiveness of the intervention, which consisted of a total of 24 sessions of 12 weeks, by making a total of two evaluations before and after the treatment.
The Loewenstein Occupational Therapy Cognitive Assessment-Geriatric (LOTCA-G) | after the 12-week intervention program
  The LOTCA-G, which was created to evaluate cognitive functions in the elderly. This test evaluates 8 cognitive domains with 24 items: orientation, visual perception, spatial perception, motor praxis, visuomotor organization, thinking operations, attention/concentration, and memory. The items in each subtest are evaluated on an ordered scale from 1 to 4 (excluding the orientation items scored from 1 to 8). A higher test score indicates better cognitive performance. The LOTCA-G can differentiate healthy older adults from those with dementia and MCI. It is sensitive to dementia levels and identifies changes over time. The LOTCA-G was used to evaluate the effectiveness of cognitive rehabilitation intervention both face-to-face and with tele-rehabilitation method. It was planned to evaluate the effectiveness of the intervention, which consisted of a total of 24 sessions of 12 weeks, by making a total of two evaluations before and after the treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Türkiye, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Torpil B, Pekcetin E, Pekcetin S. The effectiveness of cognitive rehabilitation intervention with the telerehabilitation method for amnestic mild cognitive impairment: A feasibility randomized controlled trial. J Telemed Telecare. 2025 Apr;31(3):320-327. doi: 10.1177/1357633X231189541. Epub 2023 Aug 3. PMID 37537894